CLINICAL TRIAL: NCT05134155
Title: A Pilot Study to Test the Acceptability and Feasibility of Relaxation Rooms to Help Reduce Occupational Stress Among Healthcare Workers
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Well Living Lab, Inc. (Industry)
Responsible Party: Principal Investigator, Colin West, Professor of Medicine, Mayo Clinic
Other Study IDs: 21-002545
Record Dates: First submitted 2021-11-14; First posted 2021-11-24 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Burn Out; Stress
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Test the acceptability and feasibility of a relaxation room to reduce work stress among clinicians and collect clinician-reported outcome data after using the relaxation room.

DETAILED DESCRIPTION:
The plan is to pilot test a relaxation room to demonstrate its acceptability and feasibility in the hospital and collect clinician-centered outcomes. This study will inform the design of a future trial using this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Clinician at Mayo working at St. Mary's hospital or the downtown Rochester campus during the study

Exclusion Criteria:

* Any physical condition that might prevent them from sitting for 20-30 minutes in the room
* Significant hearing loss that they would not be able to hear the audio stimuli
* Significant vision loss that they would not be able to see the visual stimuli

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Only clinicians at Mayo will be recruited as part of this study.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2022-02-26 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Acceptability | 12 months
  the proportion of clinicians who found the MindBreaks room to be somewhat acceptable or acceptable

SECONDARY OUTCOMES:
Recruitment | 12 months
  the number recruited
Room Usage | 12 months
  how long participants stayed in the MindBreaks room

CONTACTS AND LOCATIONS:
Overall Officials: Liselotte N Dyrbye, MD, MHPE, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials